CLINICAL TRIAL: NCT07064928
Title: We Are Together (WAT): Development and Testing of an Intervention to Reduce HIV Related Stigma Among Pregnant and Postpartum Women
Brief Title: Intervention to Reduce HIV Related Stigma Among Pregnant and Postpartum Women
Acronym: WAT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Africa Interdisciplinary Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01TW012893-01 (NIH); 1R01TW012893-01 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: HIV; HIV - Human Immunodeficiency Virus; Postpartum; Pregnancy; Mental Health (Depression); Mental Health; Depression - Major Depressive Disorder; Stigma; Stigma, Social; Pyschological Distress
Keywords: stigma; hiv; self stigma; anticipated stigma; enacted stigma; stigma interventions; therapy; counseling; peer interventions; postpartum women; pregnant women; women living with HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Well-Being; Depression; Social Stigma

STUDY DESIGN:
Intervention Model Description: Investigators will randomize 90 pregnant women 1:1 to intervention or standard care controls to assess F&A of the intervention and preliminary impact on outcomes. Our primary outcomes are anticipated and internalized HIV-related stigma. Secondary outcomes include ART adherence and mental health symptoms of anxiety and depression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Project Accept PTSS Module (Experimental): The adapted Project Accept's Post-Test Support Services (PTSS) Module 3 specifically designed to reduce HIV-related stigma, encourage HIV treatment adherence, and improve quality of life among those living with HIV.
  Interventions: Behavioral: Adapted Project Accept's Post-Test Support Services (PTSS) Module 3

INTERVENTIONS:
Behavioral: Adapted Project Accept's Post-Test Support Services (PTSS) Module 3 — Adapted Project Accept's Post-Test Support Services (PTSS) Module 3 for the Ghanaian context, and among pregnant and/or postpartum women living with HIV

SUMMARY:
Purpose of this Study:

The main purpose of this study is to adapt an existing evidence-based intervention, Project Accept Post-Test Support Services (PTSS) Module 3, specifically for pregnant and postpartum women living with HIV (WLWH) in Ghana. The adapted intervention aims to reduce HIV-related stigma and improve adherence to antiretroviral therapy (ART) and mental health symptoms, such as depression and anxiety, among this vulnerable population.

Why was this study done? (Background):

HIV-related stigma is a major obstacle for women living with HIV, particularly pregnant women in Sub-Saharan Africa (SSA), hindering their engagement in HIV care and adherence to ART. This contributes to poor health outcomes, including inadequate viral suppression, depression, and an ongoing risk of HIV transmission to their children and sexual partners. While effective HIV stigma-reduction interventions exist for the general adult population living with HIV, there is a critical lack of tailored interventions for pregnant and postpartum WLWH in SSA. This study addresses this gap by adapting a proven intervention (Project Accept PTSS Module 3), which has shown success in reducing stigma and improving outcomes in other populations, for this specific group in Ghana, where HIV-related stigma remains disproportionately high.

Who participated in this study? (Target Population):

This study will involve several groups:

Pregnant and postpartum women living with HIV: 30 women will participate in in-depth interviews to share their experiences with stigma and HIV care.

HIV care providers: 20 providers will participate in in-depth interviews to offer their perspectives on stigma and care provision.

Stakeholders: This group will include HIV care providers, program administrators/directors, and pregnant and postpartum women. They will collaborate in the iterative process of adapting the intervention.

Pregnant women living with HIV (for feasibility testing): 90 pregnant women will be randomized, with half receiving the adapted intervention and half receiving standard care, to assess the intervention's feasibility, acceptability, and preliminary impact.

What happened in this study? (Intervention/Methods):

This 3-year study has three main aims:

Understanding Stigma Experiences: Researchers will describe the experiences of stigma and HIV care from the perspectives of pregnant and postpartum WLWH and compare them with providers' experiences. This will involve longitudinal data collection and in-depth interviews to understand how stigma affects women's health, clinical care (e.g., provider discrimination, ART adherence), and mental health over time.

Intervention Adaptation: Project Accept PTSS Module 3 will be adapted specifically for pregnant and postpartum WLWH using the ADAPT-ITT framework. This involves an iterative process with stakeholders to ensure the intervention is culturally and gender-appropriate, enhancing its acceptability for the target population.

Feasibility and Preliminary Impact Assessment: The study will assess the feasibility and acceptability of the adapted intervention. Ninety pregnant women will be randomly assigned to either receive the intervention or continue with standard care. Researchers will then estimate the intervention's potential impact on anticipated and internalized HIV-related stigma (primary outcomes), as well as ART adherence and symptoms of anxiety and depression (secondary outcomes).

What were the results of this study? (Outcomes):

As a preliminary and adaptation study, this research aims to:

Provide essential data to inform and justify a larger, fully-powered randomized clinical trial to rigorously evaluate the adapted intervention's effectiveness.

Identify potential indicators associated with mother-to-child transmission of HIV.

Develop a model that can be applied to other Sub-Saharan African countries facing similar challenges.

Foster new collaborations focused on HIV-related stigma among women in Ghana. Build research capacity among researchers in sub-Saharan Africa.

What are the side effects of the treatments in this study? (Safety):

This study focuses on a behavioral intervention (a support and counseling module) rather than a drug or medical treatment. Therefore, typical physical side effects associated with medications are not expected. The intervention aims to improve well-being and health outcomes by addressing psychosocial factors. Any adverse events or discomfort experienced by participants will be carefully monitored and addressed in accordance with ethical guidelines.

What are the conclusions of this study? (Implications/Future Plans):

The findings from this study are expected to demonstrate the feasibility and potential impact of a culturally and gender-tailored HIV stigma-reduction intervention for pregnant and postpartum WLWH in Ghana. This research will be foundational for launching a larger-scale clinical trial to definitively test the intervention's efficacy.

DETAILED DESCRIPTION:
HIV-related stigma is a significant barrier to engagement in HIV care and adherence to antiretroviral therapy (ART), contributing to the ongoing global HIV epidemic. Stigma is a pervasive social experience in which people with marginalized attributes or identities are seen as having low social value and experience prejudice and discrimination. Globally, HIV-related stigma affects women more than men, and HIV-positive childbearing women experience even more intense stigma. In low-resource societies, pregnant women are often the first family members to receive HIV testing, a mandatory test during prenatal care, and are thus blamed and stigmatized for ostensibly bringing HIV into the family. HIV-related stigma in pregnant women also has adverse effects on infants and sero-discordant male sexual partners, who are at risk of HIV when stigma compromises the mother's ability to adhere to ART. HIV-related stigma is common in sub-Saharan Africa (SSA) where pregnant women have high HIV infection rates. HIV prevalence among women of childbearing age is increasing and this segment of the population is twice as likely to be HIV-positive than men of similar age. In SSA, HIV-related stigma among pregnant women results in poor care engagement, significant loss to follow-up, poor ART adherence, inadequate viral suppression, and depression. There is also ongoing risk of HIV transmission to their children and sexual partners. Thus, the need for intervention is critical to reducing the HIV-related stigma experienced by pregnant women in SSA to minimize loss to follow-up care and advance long-term efforts to successfully eliminate mother-to-child HIV transmission.

Prior evidence-based interventions for HIV stigma-reduction have focused on adults in the general population living with HIV but there is an absence of interventions to specifically reduce HIV stigma for pregnant and postpartum women living with HIV (WLWH) in SSA. One efficacious intervention designed for the general population is Project Accept, a US-designed multi-level intervention that significantly increased HIV testing and improved HIV outcomes. Project Accept's Post-Test Support Services (PTSS) Module 3 is specifically designed to reduce HIV-related stigma, encourage HIV treatment adherence, and improve quality of life among adults living with HIV. Participants in the United States (US) randomized to receive this module felt less stigmatized and had better ART adherence, higher retention in care, and improved well-being. The PTSS module was adapted for use in Tanzania, Nepal, South Africa and Thailand, where it led to a significant reduction in HIV-related stigma in the general population. Importantly, pregnant and postpartum WLWH were excluded from these studies.

To overcome this major gap, the investigators propose to adapt the Project Accept PTSS Module 3 specifically for pregnant and postpartum WLWH to reduce stigma and improve ART adherence and mental health symptoms of depression and anxiety. We selected Ghana in SSA for this research, where over 200,000 pregnant WLWH are placed on ART annually. While Ghana has one of the lowest HIV prevalence rates (2.3%) in SSA, the prevalence of HIV-related stigma is disproportionately high and a vast majority (≥85%) of adults express negative attitudes towards people living with HIV. The proposed intervention will be gender- and culturally-tailored to address HIV-related stigma and downstream effects on ART adherence and mental health. Our team is highly experienced in developing and testing behavioral interventions, and is conducting HIV-related stigma research in other countries within SSA. Our research aims to:

Aim 1: Describe experiences of stigma and HIV care for pregnant and postpartum WLWH compared with providers' experiences. Longitudinal data from pre- to post-natal periods and template analysis will be used to better understand women's perceptions of stigma over time and how it affects their health and clinical care (e.g., provider-based discrimination, experience of being pregnant and postpartum, mental health symptoms, adherence to ART, and HIV care engagement). The investigators will explore cultural and gender dimensions of stigma to inform the PTSS module adaptation and triangulate patient interview data (n=30) with data from providers (n=20) who will participate in in-depth interviews on their perspectives of HIV-related stigma, care provision in the context of stigma, and intervention needs.

Aim 2: Adapt Project Accept PTSS Module 3 to focus on HIV-related stigma, ART adherence, and mental health among pregnant and postpartum WLWH. Using the ADAPT-ITT framework, investigators will engage stakeholders including 1) HIV care providers, 2) program administrators/directors, and 3) pregnant and postpartum women in an iterative process of co-adapting PTSS to this population in order to establish cultural- and gender-saliency to increase the acceptability of the adapted intervention.

Aim 3: Assess feasibility and acceptability (F&A) of the intervention and estimate the potential impact on HIV-related stigma among pregnant and postpartum WLWH. Investigators will randomize 90 pregnant women 1:1 to intervention or standard care controls to assess F&A of the intervention and preliminary impact on outcomes. Our primary outcomes are anticipated and internalized HIV-related stigma. Secondary outcomes include ART adherence and mental health symptoms of anxiety and depression.

Overall Potential Impact: Results from this modular 3-year R01 will: 1) provide data needed to inform and justify a fully-powered randomized clinical trial to rigorously evaluate the adapted intervention for HIV-related stigma in pregnant and postpartum WLWH; 2) identify potential indicators associated with mother-to-child transmission of HIV; 3) serve as an applicable model for other SSA countries; 4) foster new collaborations focused on HIV-related stigma among women in Ghana; and 5) build capacity among researchers in SSA.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with HIV
* Between 24-36 weeks gestation at enrollment
* Willing to participate during the postpartum period

Recruitment process:

* Approached during a prenatal visit by a nurse/midwife
* Interested women will be connected with a trained research assistant (RA)
* RA will explain the study to potential participants

Exclusion criteria:

* Critically ill and hospitalized pregnant WLWH
* Pregnant WLWH not planning to live in the region for at least 6 months after childbirth
* Pregnant WLWH under 13 years old, under parental supervision, and attending mandatory school

Eligibility of healthcare providers:

* All providers at the four sites invited to a session at their site
* Providers eligible if they have worked with WLWH or pregnant/postpartum women for at least 2 months
* Providers who do not consent to be interviewed will not be included

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who are pregnant and/or postpartum living with HIV as identified in the local Ghanian context.
Enrollment: 175 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in anticipated HIV-related scale score | Baseline and 12 weeks
  Anticipated HIV-related stigma will be measured using Anticipated stigma scale. Response options range from 0-36 with higher scores indicating greater anticipated stigma.
Mean change in internalized HIV-related scale score | Baseline and 12 weeks
  Internalized HIV-related stigma will be measured using 10 items Internalized Stigma Scale (ISAT). Response options range from 10-50 with higher scores indicating greater internalized stigma

SECONDARY OUTCOMES:
Mean change in Edinburgh Postnatal Depression Scale (EPDS) score | Baseline and 12 weeks
  Postnatal Depression will be measured using Edinburgh Postnatal Depression Scale (EPDS). Response options range from 0-30 with higher scores indicating greater internalized stigma
Mean change in Center for Support Evaluation (CASE) scale score | Baseline and 12 weeks
  Self-report adherence will be estimated with the Center for Support Evaluation (CASE), Scores range from 3-16, and an index score of 10 or less indicates suboptimal adherence.
Presence or Absence of tenofovir (TFV) in Urine | Baseline and 12 weeks
  Point-of-care rapid test to assess tenofovir (TFV) adherence in urine will used and an immunoassay cutoff of 1500 ng/mL will classify participants as adherent. Responses will be dichotomized to "adherent/ non-adherent"

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J Ouner, PhD, RN, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Ashaiman Polyclinic, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakimuli-Mpungu E, Okello J, Kinyanda E, Alderman S, Nakku J, Alderman JS, Pavia A, Adaku A, Allden K, Musisi S. The impact of group counseling on depression, post-traumatic stress and function outcomes: a prospective comparison study in the Peter C. Alderman trauma clinics in northern Uganda. J Affect Disord. 2013 Oct;151(1):78-84. doi: 10.1016/j.jad.2013.05.055. Epub 2013 Jun 17. PMID 23787406
- [Background] Uthman OA, Magidson JF, Safren SA, Nachega JB. Depression and adherence to antiretroviral therapy in low-, middle- and high-income countries: a systematic review and meta-analysis. Curr HIV/AIDS Rep. 2014 Sep;11(3):291-307. doi: 10.1007/s11904-014-0220-1. PMID 25038748
- [Background] Sakyi KS, Lartey MY, Kennedy CE, Denison JA, Sacks E, Owusu PG, Hurley EA, Mullany LC, Surkan PJ. Stigma toward small babies and their mothers in Ghana: A study of the experiences of postpartum women living with HIV. PLoS One. 2020 Oct 16;15(10):e0239310. doi: 10.1371/journal.pone.0239310. eCollection 2020. PMID 33064737
- [Background] Khumalo-Sakutukwa G, Morin SF, Fritz K, Charlebois ED, van Rooyen H, Chingono A, Modiba P, Mrumbi K, Visrutaratna S, Singh B, Sweat M, Celentano DD, Coates TJ; NIMH Project Accept Study Team. Project Accept (HPTN 043): a community-based intervention to reduce HIV incidence in populations at risk for HIV in sub-Saharan Africa and Thailand. J Acquir Immune Defic Syndr. 2008 Dec 1;49(4):422-31. doi: 10.1097/QAI.0b013e31818a6cb5. PMID 18931624
- [Background] Coates TJ, Kulich M, Celentano DD, Zelaya CE, Chariyalertsak S, Chingono A, Gray G, Mbwambo JK, Morin SF, Richter L, Sweat M, van Rooyen H, McGrath N, Fiamma A, Laeyendecker O, Piwowar-Manning E, Szekeres G, Donnell D, Eshleman SH; NIMH Project Accept (HPTN 043) study team. Effect of community-based voluntary counselling and testing on HIV incidence and social and behavioural outcomes (NIMH Project Accept; HPTN 043): a cluster-randomised trial. Lancet Glob Health. 2014 May;2(5):e267-77. doi: 10.1016/S2214-109X(14)70032-4. Epub 2014 Apr 8. PMID 25103167
- [Background] Turan JM, Nyblade L. HIV-related stigma as a barrier to achievement of global PMTCT and maternal health goals: a review of the evidence. AIDS Behav. 2013 Sep;17(7):2528-39. doi: 10.1007/s10461-013-0446-8. PMID 23474643
- [Background] Valencia-Garcia D, Rao D, Strick L, Simoni JM. Women's experiences with HIV-related stigma from health care providers in Lima, Peru: "I would rather die than go back for care". Health Care Women Int. 2017 Feb;38(2):144-158. doi: 10.1080/07399332.2016.1217863. Epub 2016 Aug 2. PMID 27485767
- [Background] Tran BX, Phan HT, Latkin CA, Nguyen HLT, Hoang CL, Ho CSH, Ho RCM. Understanding Global HIV Stigma and Discrimination: Are Contextual Factors Sufficiently Studied? (GAPRESEARCH). Int J Environ Res Public Health. 2019 May 29;16(11):1899. doi: 10.3390/ijerph16111899. PMID 31146379
- [Background] Turan B, Stringer KL, Onono M, Bukusi EA, Weiser SD, Cohen CR, Turan JM. Linkage to HIV care, postpartum depression, and HIV-related stigma in newly diagnosed pregnant women living with HIV in Kenya: a longitudinal observational study. BMC Pregnancy Childbirth. 2014 Dec 3;14:400. doi: 10.1186/s12884-014-0400-4. PMID 25467187